CLINICAL TRIAL: NCT05045937
Title: Ivermectin Will be Used as an Outpatient Treatment Option for COVID-19 Patients.
Brief Title: Observational Study on the Use of Ivermectin as an Outpatient Treatment Option for COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Patrick Robinson (Other)
Responsible Party: Sponsor-Investigator, Patrick Robinson, Chief Investigator, Patrick Robinson MD LLC
Organization: Patrick Robinson MD LLC (Other)
Other Study IDs: Ivermectin Treatment Study #1
Record Dates: First submitted 2021-09-14; First posted 2021-09-16 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Covid19; COVID-19 Pneumonia; COVID-19 Respiratory Infection; COVID-19 Acute Bronchitis
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Ascorbic Acid; Vitamin D; Quercetin; Zinc; Budesonide; Aspirin; Acetaminophen; Ibuprofen; Infusions, Intravenous; Antibodies, Monoclonal; Melatonin; Niacin; Albuterol; remdesivir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COVID-19 patients treated with Ivermectin: This group of patients will be those who requested to be treated with Ivermectin and whom have been prescribed such by different physicians. This group may or may not include those treated with Monoclonal Antibodies or Remdesivir.
  Interventions: Drug: Ivermectin
- COVID-19 patients declining Ivermectin and wanting traditional treatment: This group of patients will be those who do not request to be treated with Ivermerctin and who want to be treated with a more traditional, minimalist approach. This group may or may not include those treated with Monoclonal Antibodies or Remdesivir.

INTERVENTIONS:
Drug: Ivermectin — Ivermectin treatment of outpatients dosing at 0.4mg/kg until recovered along with supplemental treatment using a multi-modal approach.
  Other Names: Vitamin C; Vitamin D; Quercetin; Zinc; Budesonide; Aspirin; Tylenol; Ibuprofen; IV Infusion; Monoclonal Antibodies; COVID Vaccine; Melatonin; Niacin; Albuterol; Remdesivir
  Groups: COVID-19 patients treated with Ivermectin

SUMMARY:
Ivermectin is currently being utilized by a number of physicians in the local area. My objective will be to enroll these patients at the time of their evaluation for COVID-19 infection and to follow their progress through their recovery.

DETAILED DESCRIPTION:
Patients at local physician clinics as well as my own clinic will be enrolled at the time they are evaluated for having COVID-19. Patients enrollment will be voluntary and based upon their request for treatment with Ivermectin. These patients will be questioned on symptoms and the timing of those symptoms in detail. They will then be followed throughout their treatment course to evaluate their recovery experience. Detailed accounts of their symptoms and their resolution will be followed. The study patients will stop being followed when they are either admitted to the hospital or are deemed to be symptom free. Any other medications prescribed to the patients will also be tracked. Medical histories will be taken and documented to make comparisons at the end of the study. Those patients not requesting Ivermectin will also be followed for comparisons at a later date.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 12-110 years old
* Has a recently completed COVID test
* Symptomatic and seeking treatment
* Willingness to participate and have follow-up
* Able and willing to take medications and treatment suggestions from the physician

Exclusion Criteria: Lack of symptoms, uncertain of COVID-19 status, outside of age limits for treatment

* No recent COVID test results
* Asymptomatic, even if COVID positive
* Outside of acceptable age range
* Meets criteria for hospital admission
* Unwilling to participate in trial study or have follow-up

Ages: 12 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Admitted under gender at birth
Study Population: All individuals presenting to various health clinics who are COVID positive and requesting treatment. Although the primary focus is on the effectiveness of Ivermectin for treatment, those not requesting Ivermectin treatment will be followed in a separate group.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Complete recovery from COVID-19 with resolution of symptoms | 4-6 weeks per individual
  This group recovered completely from COVID-19 and remained an outpatient throughout the duration of their illness.
Admission to a hospital for further advanced treatment | 4-6 weeks per individual
  This group of patients was unable to recover at home and required hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Patrick r Robinson, MD, Principal Investigator — Patrick Robinson MD LLC
Locations (1):
- Patrick Robinson MD LLC, San Antonio, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data may be shared at a later date once compiled.

REFERENCES:
- [Background] Simsek Yavuz S, Unal S. Antiviral treatment of COVID-19. Turk J Med Sci. 2020 Apr 21;50(SI-1):611-619. doi: 10.3906/sag-2004-145. PMID 32293834
- [Background] Trivedi N, Verma A, Kumar D. Possible treatment and strategies for COVID-19: review and assessment. Eur Rev Med Pharmacol Sci. 2020 Dec;24(23):12593-12608. doi: 10.26355/eurrev_202012_24057. PMID 33336780
- [Result] Kaur H, Shekhar N, Sharma S, Sarma P, Prakash A, Medhi B. Ivermectin as a potential drug for treatment of COVID-19: an in-sync review with clinical and computational attributes. Pharmacol Rep. 2021 Jun;73(3):736-749. doi: 10.1007/s43440-020-00195-y. Epub 2021 Jan 3. PMID 33389725
- [Result] Khan MSI, Khan MSI, Debnath CR, Nath PN, Mahtab MA, Nabeka H, Matsuda S, Akbar SMF. Ivermectin Treatment May Improve the Prognosis of Patients With COVID-19. Arch Bronconeumol (Engl Ed). 2020 Dec;56(12):828-830. doi: 10.1016/j.arbres.2020.08.007. Epub 2020 Sep 24. No abstract available. PMID 33293006
- [Result] Ahmed S, Karim MM, Ross AG, Hossain MS, Clemens JD, Sumiya MK, Phru CS, Rahman M, Zaman K, Somani J, Yasmin R, Hasnat MA, Kabir A, Aziz AB, Khan WA. A five-day course of ivermectin for the treatment of COVID-19 may reduce the duration of illness. Int J Infect Dis. 2021 Feb;103:214-216. doi: 10.1016/j.ijid.2020.11.191. Epub 2020 Dec 2. PMID 33278625
- [Result] Padhy BM, Mohanty RR, Das S, Meher BR. Therapeutic potential of ivermectin as add on treatment in COVID 19: A systematic review and meta-analysis. J Pharm Pharm Sci. 2020;23:462-469. doi: 10.18433/jpps31457. PMID 33227231
- [Result] Gupta D, Sahoo AK, Singh A. Ivermectin: potential candidate for the treatment of Covid 19. Braz J Infect Dis. 2020 Jul-Aug;24(4):369-371. doi: 10.1016/j.bjid.2020.06.002. Epub 2020 Jun 28. No abstract available. PMID 32615072
- [Result] Vallejos J, Zoni R, Bangher M, Villamandos S, Bobadilla A, Plano F, Campias C, Chaparro Campias E, Achinelli F, Guglielmone HA, Ojeda J, Medina F, Farizano Salazar D, Andino G, Ruiz Diaz NE, Kawerin P, Meza E, Dellamea S, Aquino A, Flores V, Martemucci CN, Vernengo MM, Martinez SM, Segovia JE, Aguirre MG. Ivermectin to prevent hospitalizations in patients with COVID-19 (IVERCOR-COVID19): a structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Nov 24;21(1):965. doi: 10.1186/s13063-020-04813-1. PMID 33234158